CLINICAL TRIAL: NCT05637190
Title: The Effect of Expressive Art Therapy on Teacher Burnout and Stress: A Pilot Randomized Controlled Trial
Brief Title: A Pilot RCT on the Effect of ExAT on Teacher Burnout and Stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSY025
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Burnout; Stress
Keywords: Expressive Arts Therapy; Teachers; Randomized controlled trial
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expressive Arts Therapy group (Experimental): The Expressive Arts Therapy group will receive the Expressive Arts intervention via face-to-face workshops for 2 consecutive weeks (2 hours per session). there are a total of 3 batches (around 15 participants per batch) for the intervention.
  Interventions: Other: Expressive Arts Therapy group intervention
- Waitlist control group (No Intervention): The Waitlist control group will not receive any intervention during the study, but they will receive self-help art therapy materials after the whole study procedure.

INTERVENTIONS:
Other: Expressive Arts Therapy group intervention — Art is helpful to reduce negative emotions and boost self-worth during the creative process. During the Expressive Arts Therapy workshops, participants experience different art forms, including visual art, body movement, writing, music, and guided imagery to identify the inner self and get in touch with the self to release suppressed emotions and stress.
  Arms: Expressive Arts Therapy group

SUMMARY:
The objective of this pilot randomized controlled trial is to evaluate the effects of Expressive Art Therapy on reducing burnout and stress symptoms among Hong Kong's primary and secondary school teachers.

The proposed study is a pilot randomized controlled trial. Prior to all study procedures, 90 participants (i.e., primary and secondary school teachers) will be recruited to complete an online informed consent with telephone support. Eligible participants will be randomly assigned to either the Expressive Arts Therapy group (ExAT group) or the waitlist control group (WL group) in a ratio of 1:1. The ExAT group will receive the Expressive Arts intervention via face-to-face workshops for 2 consecutive weeks (2 hours per session). There are a total of 3 batches (around 15 participants per batch) for the intervention. Participants in this group will be in touch with their inner selves and inner resources via body movement, writing and music. There will be visual art creation as a conclusion for integrating the body and mind. The art products would be placed in their workplace for stress regulation. The WL control group will not receive any intervention during the study, but they will receive self-help art therapy materials after the whole study procedure. The outcome measures include burnout, stress, depressive, and anxiety symptoms, as well as insomnia symptoms, physical activity, health-related quality of life, and the intervention acceptability at baseline, immediate post-treatment, and 4-week follow-up assessments by completing the same questionnaire set.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged >/=18
2. Able to read Chinese (verbal expression in Chinese or English)
3. With qualified teaching cert. (degree holder)
4. Willing to provide informed consent and comply with the trial protocol
5. Teacher work in primary or secondary school in Hong Kong

Exclusion Criteria:

1. Current involvement in psychological treatment program for stress and / or burnout reduction
2. A change in psychotropic drugs or over-the-counter medications that target mood within 2 weeks before the baseline assessment
3. A Patient Health Questionnair-9 (PHQ-9) item 9 score > 2 indicating a serious level of suicidal risk

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Shirom-Melamed Burnout Measure (SMBM) | baseline (week 0), immediate post intervention (week 3) and 4-week post intervention follow up
  A 14-item questionnaire with 7-point scale will be used for physical fatigue, emotion exhaustion, and cognitive weariness. The score ranges from 1(never or almost never) to 7 (always or almost always). Item 1-5: physical fatigue; item 6-8: emotional exhaustion; and item 9-14: cognitive wariness
Change in Perceived Stress Scale (PSS) | baseline (week 0), immediate post intervention (week 3) and 4-week post intervention follow up
  A 10-item questionnaire measuring the perceived degree of stress across situations over the past month. Items include how unpredictable, uncontrollable, and overloaded do the respondents perceive. the score ranges from 0 (never) to 4 (very often)

SECONDARY OUTCOMES:
Change in The Patient Health Questionnaire (PHQ-9) | baseline (week 0), immediate post intervention (week 3) and 4-week post intervention follow up
  A 9-item questionnaire used for screening, diagnosing, monitoring, and measuring the severity of depression, which scores each of the nine DSM-IV criteria as 0 (not at all) to 3 (nearly every day)
Change in The Generalized Anxiety disorder 7-item Scale (GAD-7) | baseline (week 0), immediate post intervention (week 3) and 4-week post intervention follow up
  A brief 7-item instrument for screening for generalized anxiety disorder and assessing its severity in clinical practice and research. Anxiety severity is categorized using scores of 5-9 (mild), 10-14 (moderate) and 15or more (severe)
Change in Insomnia Severity Index (ISI) | baseline (week 0), immediate post intervention (week 3) and 4-week post intervention follow up
  A 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem and level of distress caused by the sleep problem.
Change in Multidimensional Fatigue Inventory (MFI-20) | baseline (week 0), immediate post intervention (week 3) and 4-week post intervention follow up
  A 20-item self-report instrument designed to measure fatigue. Ratings on a 5-point Likert sscale are obtained on the dimensions of general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. Scores on each subscale range from 4 to 20, with higher scores indicating greater fatigue
Change in Short Form (Six-Dimension) Health Survey - The Chinese (Hong Kong) Version (SF-6D) | baseline (week 0), immediate post intervention (week 3) and 4-week post intervention follow up
  A preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health and vitality. The SF-6D index, scored from 0.0 (worst health state) to 1.0 (best health state)
Change in Credibility-Expectancy questionnaire (CEQ) | baseline (week 0), immediate post intervention (week 3) and 4-week post intervention follow up
  The 6-item CEQ yielded ratings of treatement credibility, acceptability/satisfaction, and expectations for success
Change in Treatment Acceptability and Adherence Scale (TAAS) | baseline (week 0), immediate post intervention (week 3) and 4-week post intervention follow up
  A 10-item self-report scale designed to measure treatment acceptability on various facets, such as dropout likelihood and treatment adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona YY Ho, Ph.D, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No